CLINICAL TRIAL: NCT05259787
Title: Efficacy and Safety of Etomidate Combined with Propofol Intravenous Anesthesia During Hysteroscopic Procedures: a Randomized Controlled Trial
Brief Title: EP Intravenous Anesthesia in Hysteroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP hysteroscopy
Record Dates: First submitted 2021-12-20; First posted 2022-03-02 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia
Keywords: propofol; etomidate; intravenous anesthesia; hysteroscopic surgery
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etomidate combined with propofol（EP） (Experimental): 0.2ml/kg IV
  Interventions: Drug: Sedation Etomidate combined with propofol
- Propofol（P） (Active Comparator): 0.2ml/kg IV
  Interventions: Drug: Sedation Propofol

INTERVENTIONS:
Drug: Sedation Etomidate combined with propofol — Drug IV within 10 second during anesthesia induction.
  Other Names: EP
  Arms: Etomidate combined with propofol（EP）
Drug: Sedation Propofol — Drug IV within 10 second during anesthesia induction.
  Other Names: EP
  Arms: Propofol（P）

SUMMARY:
Hysteroscopy is a gold standard method for evaluating the uterine cavity and diseases, which is gradually becoming a day-surgery in China. Propofol is one of the most commonly used intravenous anesthetics in clinic for hysteroscopic procedures, however high dose propofol bring some potential clinical safety hazards.In this study, the feasibility and safety of Etomidate combined with propofol(1:2) as improved scheme for hysteroscopic surgery will be evaluated.

DETAILED DESCRIPTION:
Hysteroscopy is a gold standard method for evaluating the uterine cavity and diseases, which is gradually becoming a day-surgery in China. For hysteroscopic surgery using bipolar resectoscopes, hysteroscopic morcellators or shavers, it is considered efficient and safe to be performed under general anaesthesia, such as intravenous anesthesia. Propofol is one of the most commonly used intravenous anesthetics in clinic, however high dose propofol bring some potential clinical safety hazards, reducing respiratory rate and tidal volume, causing apnea or hypoxemia, and leading to hypoxia especially for obese and elderly patients. Propofol combined with etomidate as an improved scheme of intravenous anesthesia has been proved to have advantages in gastroendoscopy.In this study, the patients undergoing elective hysteroscopic surgery will be randomly assigned to two groups of intravenous anesthesia: Etomidate combined with propofol of 1:2 ratio (EP) versus Propofol (P). The sedation degree, respiratory related events (hypoxia, asphyxia incidence and maintenance time) and hemodynamic events，integrated pulmonary index (IPI) of the two groups will be evaluated to explore the feasibility and safety of the clinical application of EP mixture in hysteroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective hysteroscopic surgery;
* intravenous anesthesia;
* normal reading and understanding ability
* volunteer to participate

Exclusion Criteria:

* serious complications such as heart failure, liver failure, pulmonary dysfunction, renal failure, etc.
* predictable difficult airway
* high risk of reflux aspiration
* allergy to propofol or etomidate
* already participated in other clinical trials within three months before admission
* unwilling to cooperate

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Modified observer's assessment of alert /sedation scores (MOAAS scores) | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Modified observer's assessment of alert /sedation score 0-2 as effective anesthesia for hysteroscopic procedures.The MOAAS scores is a 6-point scale that assesses the responsiveness of patients and coincides with the ASA continuum of sedation. A patient with a score of 5 responds readily to name spoken in a normal tone, 4 lethargic response to name spoken in a normal tone, 3 responds only after the name is called loudly and/or repeatedly, 2 responds only after mild prodding or shaking, 1 responds only after painful trapezius squeeze, and 0 does not respond to painful trapezius squeeze (0 to 1 deep sedation, 2 to 4 moderate sedation, and 5 minimal sedation or alert).
Apnea duration | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  The time duration from the disappearance to the recovery of spontaneous breathing, record in seconds.

SECONDARY OUTCOMES:
Incidence of manual ventilation intervention | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  When Pulse Oxygen Saturation(SpO2)<90% ，mask pressure ventilation or mechanical ventilation should be used as the intervention. The intervention incidence will be record in percentage.
Pulse oxygen saturation (SpO2) | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Pulse oxygen saturation (SpO2) will be recorded in percentage, range from 0 to 100%.
Blood Pressure(BP) | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Noninvasive blood pressure will be recorded in mmHg.
Heart rate (HR) | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Heart rate (HR) will be recorded in times/min.

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, MD,PHD, Study Director — Renji Hospital, Shanghai Jiaotong University, School of Medcine
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No